CLINICAL TRIAL: NCT05697055
Title: A Prospective Multicenter, Randomized, Controlled Clinical Trial of the Safety and Efficacy of Azvudine vs. Nirmatrelvir-Ritonavir in Hospitalized Patients With Moderate to Severe COVID-19 Infection
Brief Title: A Study of Efficacy and Safety of Azvudine vs. Nirmatrelvir-Ritonavir in the Treatment of COVID-19 Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Collaborators: Qianfoshan Hospital (Other); The Second Affiliated Hospital of Shandong First Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); Gansu Provincial Hospital (Other); Rizhao People's Hospital (Other)
Responsible Party: Principal Investigator, Jia-jun Zhao, Director, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWYX2023022
Record Dates: First submitted 2023-01-20; First posted 2023-01-25 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: COVID-19; Azvudine; Nirmatrelvir-Ritonavir; Efficacy; Safety
MeSH Terms: conditions — COVID-19 | interventions — azvudine; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azvudine (Experimental)
  Interventions: Drug: Azvudine
- Nirmatrelvir-Ritonavir (Active Comparator)
  Interventions: Drug: Nirmatrelvir-Ritonavir

INTERVENTIONS:
Drug: Azvudine — 5mg orally, once a day, for no more than 14 days
  Arms: Azvudine
Drug: Nirmatrelvir-Ritonavir — Nirmatrelvir 300mg combined with Ritonavir 100mg every 12 hours for 5 days. For patients with 30≤ eGFR < 60 ml/min, it should be reduced to150mg/100mg Nirmatrelvir-Ritonavir every 12 hours for 5 days
  Arms: Nirmatrelvir-Ritonavir

SUMMARY:
The COVID-19 pandemic has become a major public health challenge, and the treatment options for the disease are currently limited. The commonly used oral small-molecule anti-COVID-19 drugs in China are Nirmatrelvir-Ritonavir and Azvudine. These drugs have been tested in pre-marketing clinical trials in patients with non-severe COVID-19 infection and have demonstrated therapeutic effects in inhibiting virus transmission and preventing disease progression. However, until now, the efficacy and safety of these drugs in patients with moderate to severe COVID-19 infections remains unclear. Therefore, this study is aiming to compare the efficacy and safety of Azvudine and Nirmatrelvir-Ritonavir in moderate to severe COVID-19 infections. This study will be a multicenter, randomized, controlled clinical trial study in patients hospitalized with moderate to severe COVID-19 infections. Recovery of clinical symptoms, nucleic acid negative conversion, improvement in oxygenation index, and imaging improvement will be used as study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients of ≥18 years old, regardless of gender or race;
2. Patients who have a positive SARS-CoV-2 test result;
3. Diagnosed with moderate or severe COVID-19 infection according to the diagnostic criteria from the "Diagnosis and treatment program trial version 10 guidelines" issued by the National Health Commission of the People's Republic of China. Including:

   ①Moderate: continuous high fever for more than 3 days or/and cough, shortness of breath, etc., but the breathing frequency (RR) is less than 30 times/minute, and the oxygen saturation when inhaling air at rest is > 93%. Imaging shows the characteristic manifestations of COVID-19 pneumonia.

   ② Severe: Adults meet any of the following requirements: A, shortness of breath, RR≥ 30 times/minute; B, the oxygen saturation when inhaling air at rest is ≤ 93%; C, Arterial partial oxygen pressure (PaO2)/ Fraction of inspiration O2 (FiO2) ≤300mmHg (1mmHg=0.133kPa), and PaO2/FiO2 should be corrected according to the following formula for areas above 1000 m :PaO2/FiO2× [760/ atmospheric pressure (mmHg)]; D, the clinical symptoms were gradually aggravated, and the lung imaging showed that the lesion progressed significantly within 24 ~ 48 hours > 50%.
4. Join this study voluntarily.
5. Each subject must sign an informed consent form (ICF) indicating that he/she understands the purpose and procedure of the study and is willing to participate in the study. Considering the patient's condition, the ICF may be signed by the legal representative.

Exclusion Criteria:

1. Allergic to the drugs involved;
2. Pregnancy or lactation;
3. Diagnosed or suspected critical COVID-19 infection;
4. Child-Pugh C of liver function or estimated glomerular filtration rate (eGFR) less than 30mL/min during screening;
5. Receive SARS-CoV-2 monoclonal antibody therapy or other antiviral therapy;
6. The subject and/or authorized family members refused to receive anti-COVID-19 treatment;
7. Any life-threatening disease or organ system dysfunction that the researcher thinks can harm the safety of the subjects and expose the research results to unnecessary risks; drug addicts, uncontrolled mental illness or cognitive dysfunction.
8. Join other similar clinical researchers within 3 months;
9. Patients who were not considered suitable for inclusion by the researchers (such as patients who were expected to be unable to adhere to the treatment due to financial problems).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-05-21 (Estimated); Study Completion 2023-07-21 (Estimated)

PRIMARY OUTCOMES:
Time and proportion of patients with COVID-19 infection to have sustained clinical recovery | Up to 28 days

SECONDARY OUTCOMES:
Proportion of progression to critical COVID-19 and death from any cause | Up to 28 days
Time of COVID-19 related symptom score and World Health Organization (WHO) clinical progress scale score. Time and proportion of clinical recovery, symptom resolution and regression of major symptoms | Up to 28 days
Time and proportion of the nucleic acid negative conversion | Days 3, 6, 9, 12, 15, 18, 21, 24, 27
Time and proportion of chest CT image improvement | Days 6, 12, 18, 24
Time and proportion of oxygenation index improvement | Up to 28 days
Length of stay | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China